CLINICAL TRIAL: NCT01236560
Title: A Randomized Phase II/III Study of Vorinostat and Local Irradiation OR Temozolomide and Local Irradiation OR Bevacizumab and Local Irradiation Followed by Maintenance Bevacizumab and Temozolomide in Children With Newly Diagnosed High-Grade Gliomas
Brief Title: Vorinostat, Temozolomide, or Bevacizumab in Combination With Radiation Therapy Followed by Bevacizumab and Temozolomide in Young Patients With Newly Diagnosed High-Grade Glioma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02616; NCI-2011-02616 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000688443; ACNS0822; 11-00910; ACNS0822 (Other: Children's Oncology Group); ACNS0822 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Results first posted 2020-06-22 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Brain Stem Glioma; Cerebral Astrocytoma; Childhood Cerebellar Anaplastic Astrocytoma; Childhood Cerebral Anaplastic Astrocytoma; Childhood Spinal Cord Neoplasm
MeSH Terms: conditions — Astrocytoma; Spinal Cord Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Temozolomide; Vorinostat

ARMS (6):
- Arm I (vorinostat, Phase II Arm A) (Experimental): Patients undergo RT 5 days a week for 6 weeks and receive vorinostat at the maximum-tolerated dose determined in the feasibility study. Patients receive Maintenance therapy of bevacizumab 10mg/kg/dose every 2 weeks and temozolomide 200 mg/m2/dose Days 1-5, for up to twelve cycles in the absence of progressive disease and unacceptable toxicities.
  Interventions: Biological: Bevacizumab; Drug: Temozolomide; Drug: Vorinostat
- Arm II (temozolomide, Phase II Arm B) (Experimental): Patients undergo RT as in the feasibility arm and receive temozolomide PO once daily for 42 days by day 5 of RT. Patients receive Maintenance therapy of bevacizumab 10mg/kg/dose every 2 weeks and temozolomide 200 mg/m2/dose Days 1-5, for up to twelve cycles in the absence of progressive disease and unacceptable toxicities.
  Interventions: Biological: Bevacizumab; Drug: Temozolomide
- Arm III (Bevacizumab, Phase II Arm) (Experimental): Patients undergo RT as in the feasibility arm and receive bevacizumab IV over 30-90 minutes on days 22 and 36. Patients receive Maintenance therapy of bevacizumab 10mg/kg/dose every 2 weeks and temozolomide 200 mg/m2/dose Days 1-5, for up to twelve cycles in the absence of progressive disease and unacceptable toxicities.
  Interventions: Biological: Bevacizumab; Drug: Temozolomide
- Arm IV (temozolomide, Phase 3 Arm B) (Experimental): Patients undergo RT as in the Arm II and receive temozolomide PO once daily for 42 days beginning on day 5 of RT. Patients receive Maintenance therapy of bevacizumab 10mg/kg/dose every 2 weeks and temozolomide 200 mg/m2/dose Days 1-5, for up to twelve cycles in the absence of progressive disease and unacceptable toxicities.
  Interventions: Biological: Bevacizumab; Drug: Temozolomide
- Arm V (vorinostat/bevacizumab, Phase 3, Chemoradiotherapy) (Experimental): Patients receive treatment as in phase II, arm I or phase II, arm III, whichever was established as superior in phase II. Patients receive Maintenance therapy of bevacizumab 10mg/kg/dose every 2 weeks and temozolomide 200 mg/m2/dose Days 1-5, for up to twelve cycles in the absence of progressive disease and unacceptable toxicities.
  Interventions: Biological: Bevacizumab; Drug: Temozolomide; Drug: Vorinostat
- Feasibility (vorinostat) (Experimental): Patients undergo RT 5 days a week for 6 weeks and receive vorinostat at 230 mg/m2/day. In the event of 2 or more DLTs, participants will de-escalate to vorinostat at 180 mg/m2/day. Patients receive Maintenance therapy of bevacizumab 10mg/kg/dose every 2 weeks and temozolomide 200 mg/m2/dose Days 1-5, for up to twelve cycles in the absence of progressive disease and unacceptable toxicities.
  Interventions: Biological: Bevacizumab; Drug: Temozolomide; Drug: Vorinostat

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; CT-P16; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; MYL-1402O; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ
Drug: Vorinostat — Given PO
  Other Names: L-001079038; MSK-390; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza
  Arms: Arm I (vorinostat, Phase II Arm A); Arm V (vorinostat/bevacizumab, Phase 3, Chemoradiotherapy); Feasibility (vorinostat)

SUMMARY:
This randomized phase II/III trial is studying vorinostat, temozolomide, or bevacizumab to see how well they work compared with each other when given together with radiation therapy followed by bevacizumab and temozolomide in treating young patients with newly diagnosed high-grade glioma. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Radiation therapy uses high-energy x-rays to kill tumor cells. It is not yet known whether giving vorinostat is more effective then temozolomide or bevacizumab when given together with radiation therapy in treating glioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify the dose of vorinostat that is feasible when given in combination with radiotherapy (RT) in patients with newly diagnosed high-grade gliomas (HGG). II. To compare 1-year event-free survival of patients with newly diagnosed HGG treated with vorinostat (using MTD) versus bevacizumab versus temozolomide when given in combination with RT followed by maintenance therapy with bevacizumab and temozolomide. (Phase II) III. To compare the event-free survival of patients with newly diagnosed HGG treated with the superior chemoradiotherapy (from phase II portion) versus temozolomide given in combination with RT followed by maintenance chemotherapy with bevacizumab and temozolomide. (Phase III)

SECONDARY OBJECTIVES:

I. To evaluate the anti-tumor activity, as measured by event-free survival (EFS), progression-free survival (PFS), and overall survival (OS), of patients with newly diagnosed HGG treated with vorinostat, bevacizumab, or temozolomide when given in combination with RT followed by maintenance chemotherapy with bevacizumab and temozolomide. II. To define and evaluate the toxicities of each of the treatment arms of the study.

III. To conduct gene expression profiling and SNP arrays in patients with newly diagnosed HGG.

IV. To assess telomerase activity, hTert expression, and telomere length in patients with newly diagnosed HGG. V. To document changes in perfusion and diffusion using MR imaging at baseline, prior to, during (prior to course 3), and after maintenance therapy with bevacizumab and temozolomide.

VI. To correlate functional changes in tumor with responses to bevacizumab treatment using MR diffusion/perfusion imaging. VII. To correlate the results of the bevacizumab biology studies in serum or tumor with EFS.

VIII. To explore the prognostic significance of MGMT status for patients newly diagnosed with HGG treated with combined surgery, radiation, chemotherapy, and anti-angiogenic therapy.

OUTLINE: This is a multicenter, feasibility, dose-escalation study of vorinostat, followed by a phase II study, followed by a phase III study.

FEASIBILITY STUDY: Patients undergo 3-D conformal radiotherapy (RT) or intensity-modulated RT 5 days a week for 6 weeks. Patients also receive vorinostat orally (PO) once daily on days 1-5. Courses repeat every week for 6 weeks in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Beginning 4 weeks after completion of chemoradiotherapy, patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and temozolomide PO on days 1-5. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.

PHASE II STUDY: Patients are stratified according to extent of resection (near total resection or gross total resection vs other) and histology (glioblastoma multiforme vs other). Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients undergo RT 5 days a week for 6 weeks and receive vorinostat at the maximum-tolerated dose determined in the feasibility study.

ARM II: Patients undergo RT as in the feasibility arm and receive temozolomide PO once daily for 42 days by day 5 of RT.

ARM III: Patients undergo RT as in the feasibility arm and receive bevacizumab IV over 30-90 minutes on days 22 and 36.

Maintenance therapy in arms I, II, III: Patients in all arms receive maintenance therapy as in the feasibility study.

PHASE III study: Patients are randomized to 1 of 2 treatment arms.

ARM IV: Patients receive RT and temozolomide as in phase II, arm II.

ARM V: Patients receive treatment as in phase II, arm I or phase II, arm III, whichever was established as the superior chemoradiotherapy arm in phase II.

Maintenance Therapy: Beginning 4 weeks after completion of chemoradiotherapy, patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and temozolomide PO on days 1-5. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity. Some patients undergo blood and tumor tissue sample (from surgery) collection for telomerase activity, hTert expression, telomere length, and gene expression profiling and SNP arrays analysis.

After completion of study therapy, patients are followed up every 3 months for 1 year, every 6 months for 4 years, and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed high-grade glioma

  * Anaplastic astrocytoma
  * Glioblastomamultiforme
  * Gliosarcoma
  * Primary spinal cord malignant glioma allowed
  * No oligodendroglioma oroligoastrocytoma
* Patient must have histological verification of diagnosis

  * No M+ disease (defined as evidence of neuraxis dissemination)
  * No positive CSF cytology
* ECOG performance status (PS) 0-2

  * Karnofsky PS 50-100% (patients > 16 years of age)
  * Lansky PS 50-100% (patients ≤ 16 years of age)
* ANC ≥ 1,000/μL
* Platelet count ≥ 100,000/μL
* Hemoglobin ≥ 8.0 mg/dL (transfusion independent)
* Creatinine clearance or radioisotope GFR ≥ 70 mL/min OR serum creatinine based on age and/or gender as follows:

  * 0.4 mg/dL (1 month to < 6 months of age)
  * 0.5 mg/dL (6 months to < 1 year of age)
  * 0.6 mg/dL (1 to < 2 years of age)
  * 0.8 mg/dL (2 to < 6 years of age)
  * 1.0 mg/dL (6 to < 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 mg/dL (male) or 1.4 mg/dL (female) (13 to < 16 years of age)
  * 1.7 mg/dL (male) or 1.4 mg/dL (female) (≥ 16 years of age)
* Proteinuria < 2+ OR urine; protein ratio (UPC) ≤ 0.5

  * If UPC > 0.5, a 24-hour urine protein should be obtained and level should be < 1,000 mg of protein
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT < 2.5 times ULN
* Serum albumin ≥ 2 g/dL
* PT INR ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during all study therapy and for ≥ 6 months after completion of bevacizumab
* Hypertension well controlled (≤ 95^th percentile for age and height if patient is ≤ 17years) by stable doses of medication allowed

  * For patients > 17 years, systolic blood pressure (BP) ≤ 150 mm Hg or diastolic BP ≤ 100 mm Hg)
* Seizure disorder allowed provided patient is well-controlled and on nonenzyme-inducing anticonvulsants
* No history of myocardial infarction, severe or unstable angina, clinically significant peripheral vascular disease, ≥ grade 2 heart failure, or serious and inadequately controlled cardiac arrhythmia
* No known bleeding diathesis or coagulopathy
* No prior arterial thromboembolic events, including transient ischemic attacks orcerebrovascular accidents
* No prior diagnosis of a deep venous thrombosis, including pulmonary embolism, and no known thrombophilic condition (e.g., protein S, protein C, antithrombin III deficiency, Factor V Leiden or Factor II G202'0A mutation, homocysteinemia, or antiphospholipid antibody syndrome)
* No history of an abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No serious or non-healing wound, ulcer, or bone fracture
* No evidence of significant postoperative intracranial hemorrhage, defined as > 1 cm of blood on postoperative MRI scan (potentially in addition to the postoperative scan) obtained within the past 14days
* No history of allergic reaction to Chinese hamster ovary cell products or other recombinanthuman antibodies
* No more than 31 days since definitive surgery
* Must not have received any prior chemotherapy, radiotherapy, immunotherapy, or bone marrow transplant
* More than 7 days since major surgical procedure and recovered

  * For patients scheduled to receive bevacizumab:

    * More than 28 days since major procedure
    * More than 14 days since intermediate procedure
    * More than 7 days since minor procedure (lumbar picture or placement of PICC lines are not considered minor procedures)
* No other current anti-cancer agents
* No concurrent nonsteroidal anti-inflammatory medications known to inhibit platelet function or known to selectively inhibit cyclooxygenase activity
* No concurrent enzyme inducing anticonvulsants
* No concurrent HDAC inhibitors (e.g., valproic acid)
* No concurrent anticoagulants including systemic thrombolytic agents, heparin, low molecular weight heparins, or warfarin except as required to maintain patency of pre-existing permanent vascular catheters or for prevention of thrombosis in the post-operative period

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 101 (Actual)
Dates: Start 2011-01-26 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Fouladi, Principal Investigator — Children's Oncology Group
Locations (132):
- United States (124):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Oncology Group, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (8):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After one-year EFS, neither Vorinostat nor Bevacizumab were found superior to temozolomide, therefore Phase III portion of the study did not occur.
Groups:
- Arm III (Bevacizumab, Phase II Arm C): Patients undergo RT as in the feasibility arm and receive bevacizumab IV over 30-90 minutes on days 22 and 36. Patients receive Maintenance therapy of bevacizumab 10mg/kg/dose every 2 weeks and temozolomide 200 mg/m2/dose Days 1-5, for up to twelve cycles in the absence of progressive disease and unacceptable toxicities.
  Bevacizumab: Given IV
  Temozolomide: Given PO
- Arm IV (Temozolomide, Phase III Arm B): Patients undergo RT as in the Arm II and receive temozolomide PO once daily for 42 days beginning on day 5 of RT. Patients receive Maintenance therapy of bevacizumab 10mg/kg/dose every 2 weeks and temozolomide 200 mg/m2/dose Days 1-5, for up to twelve cycles in the absence of progressive disease and unacceptable toxicities.
  Bevacizumab: Given IV
  Temozolomide: Given PO
- Arm V (Vorinostat/Bevacizumab, Phase III, Chemoradiotherapy: Patients receive treatment as in phase II, arm I or phase II, arm III, whichever was established as superior in phase II. Patients receive Maintenance therapy of bevacizumab 10mg/kg/dose every 2 weeks and temozolomide 200 mg/m2/dose Days 1-5, for up to twelve cycles in the absence of progressive disease and unacceptable toxicities.
  Bevacizumab: Given IV
  Temozolomide: Given PO
  Vorinostat: Given PO
Period: Overall Study
Arm/Group | Feasibility (Vorinostat) | Arm I (Vorinostat, Phase II Arm A) | Arm II (Temozolomide, Phase II Arm B) | Arm III (Bevacizumab, Phase II Arm C) | Arm IV (Temozolomide, Phase III Arm B) | Arm V (Vorinostat/Bevacizumab, Phase III, Chemoradiotherapy
Started | 6 | 32 | 31 | 32 | 0 | 0
Completed | 1 | 8 | 11 | 10 | 0 | 0
Not Completed | 5 | 24 | 20 | 22 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 1 | 3 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 8 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Progressive disease | 5 | 19 | 9 | 16 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Since neither Vorinostat nor Bevacizumab were found superior to temozolomide, there were no patients to analyze for Phase III
Groups:
- Total: Total of all reporting groups
Arm/Group | Feasibility (Vorinostat) | Arm I (Vorinostat, Phase II Arm A) | Arm II (Temozolomide, Phase II Arm B) | Arm III (Bevacizumab, Phase II Arm C) | Arm IV (Temozolomide, Phase III Arm B) | Arm V (Vorinostat/Bevacizumab, Phase III, Chemoradiotherapy | Total
Number analyzed (Participants) | 6 | 32 | 31 | 32 | 0 | 0 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 29 | 29 | 29 | 0 | 0 | 93
  Between 18 and 65 years | 0 | 3 | 2 | 3 | 0 | 0 | 8
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 12.6 [9.7 to 15.5] | 12.2 [4.1 to 20.7] | 11.3 [3.7 to 22.0] | 11.8 [3.4 to 20.0] |  |  | 11.8 [3.4 to 22.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 16 | 15 | 12 | 0 | 0 | 46
  Male | 3 | 16 | 16 | 20 | 0 | 0 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 6 | 3 | 0 | 0 | 13
  Not Hispanic or Latino | 6 | 26 | 24 | 27 | 0 | 0 | 83
  Unknown or Not Reported | 0 | 2 | 1 | 2 | 0 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 1 | 1 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 6 | 3 | 0 | 0 | 9
  White | 6 | 25 | 21 | 27 | 0 | 0 | 79
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 2 | 1 | 0 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Vorinostat
Description: The dose of vorinostat in mg/sq m/day to be administered with combination chemotherapy and radiation therapy.
Time Frame: 10 weeks
Population: MTD is determined using only patients treated with vorinostat
Measure: Number; unit: mg/sq m
Arm/Group | Feasibility (Vorinostat)
Number analyzed (Participants) | 6
mg/sq m | 230

2. Primary Outcome: Event-free Survival
Description: Time from enrollment to disease progression, diagnosis of a second malignant neoplasm, death or last follow-up, whichever occurs first. Disease progression is evaluated according to the COG criteria for measurement of brain tumors and is defined to be a ≥ 25% increase in the product of perpendicular diameters of ANY target lesion, taking as reference the smallest product observed since the start of treatment; OR the appearance of one or more new lesions, OR worsening neurologic status not explained by causes unrelated to tumor progression (e.g., anticonvulsant or corticosteroid toxicity, electrolyte disturbances, sepsis, hyperglycemia, presumed post-therapy swelling etc) PLUS any increase in tumor cross-sectional area (or tumor volume).
Time Frame: 1 year after enrollment
Population: Only eligible patients included in analysis
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Feasibility (Vorinostat) | Arm I (Vorinostat, Phase II Arm A) | Arm II (Temozolomide, Phase II Arm B) | Arm III (Bevacizumab, Phase II Arm C)
Number analyzed (Participants) | 6 | 31 | 27 | 32
percent probability | 33.3 [26.6 to 68] | 41.3 [23.7 to 58.3] | 59.3 [38.6 to 75.0] | 43.8 [26.5 to 59.8]

3. Secondary Outcome: Overall Survival
Description: Time from enrollment to death or last follow-up, whichever occurs first.
Time Frame: 1 year after enrollment
Population: Only eligible patients included in analysis
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Feasibility (Vorinostat) | Arm I (Vorinostat, Phase II Arm A) | Arm II (Temozolomide, Phase II Arm B) | Arm III (Bevacizumab, Phase II Arm C)
Number analyzed (Participants) | 6 | 31 | 27 | 32
percent probability | 33.3 [2.6 to 68] | 82.2 [62.5 to 92.2] | 85.2 [65.2 to 94.2] | 67.3 [47.7 to 80.9]

4. Secondary Outcome: Cumulative Incidence of Disease Progression in Each Treatment Arm
Description: Cumulative incidence of progression where death from any cause prior to progression and diagnosis of a second malignant neoplasm prior to progression are considered competing events. Disease progression is evaluated according to the COG criteria for measurement of brain tumors and is defined to be a ≥ 25% increase in the product of perpendicular diameters of ANY target lesion, taking as reference the smallest product observed since the start of treatment; OR the appearance of one or more new lesions, OR worsening neurologic status not explained by causes unrelated to tumor progression (e.g., anticonvulsant or corticosteroid toxicity, electrolyte disturbances, sepsis, hyperglycemia, presumed post-therapy swelling etc) PLUS any increase in tumor cross-sectional area (or tumor volume).
Time Frame: 1 year after enrollment
Population: Only eligible patients included in analysis.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Feasibility (Vorinostat) | Arm I (Vorinostat, Phase II Arm A) | Arm II (Temozolomide, Phase II Arm B) | Arm III (Bevacizumab, Phase II Arm C)
Number analyzed (Participants) | 6 | 31 | 27 | 32
percent probability | 67 [22 to 100] | 59 [40 to 77] | 53 [35 to 71] | 37 [18 to 56]

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution, via expedited reporting (NCI AdEERs / CAeRs). The "AE Other" table reflects all CTCAEs collected excluding those that were reported as SAEs. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Feasibility (Vorinostat) | Arm I (Vorinostat, Phase II Arm A) | Arm II (Temozolomide, Phase II Arm B) | Arm III (Bevacizumab, Phase II Arm C)
All-Cause Mortality (participants affected / at risk) | 5/6 | 24/29 | 22/27 | 23/32
Serious Adverse Events (participants affected / at risk) | 4/6 | 9/29 | 10/27 | 12/32
Other Adverse Events (participants affected / at risk) | 2/6 | 13/29 | 14/27 | 16/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Feasibility (Vorinostat) (N=6) | Arm I (Vorinostat, Phase II Arm A) (N=29) | Arm II (Temozolomide, Phase II Arm B) (N=27) | Arm III (Bevacizumab, Phase II Arm C) (N=32)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Optic nerve disorder (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 0 (0) | 3 (3) | 5 (5) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Hydrocephalus (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Feasibility (Vorinostat) (N=6) | Arm I (Vorinostat, Phase II Arm A) (N=29) | Arm II (Temozolomide, Phase II Arm B) (N=27) | Arm III (Bevacizumab, Phase II Arm C) (N=32)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 3 (3) | 3 (3) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (3) | 5 (5) | 8 (8)
Platelet count decreased (Investigations) | 0 (0) | 5 (5) | 8 (8) | 6 (6)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 2 (2) | 5 (5) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-12-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT01236560/Prot_SAP_000.pdf